CLINICAL TRIAL: NCT03423628
Title: A Phase I, Multicenter Study to Assess the Safety, Tolerability, and Pharmacokinetics of Ascending Doses of AZD1390 in Combination With Radiation Therapy in Patients With Glioblastoma Multiforme and Brain Metastases From Solid Tumors
Brief Title: A Study to Assess the Safety and Tolerability of AZD1390 Given With Radiation Therapy in Patients With Brain Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6940C00002; 135803 (Registry Identifier: IND); 2017-002451-28 (EudraCT Number)
Record Dates: First submitted 2017-11-28; First posted 2018-02-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Glioblastoma Multiforme; Primary Glioblastoma Multiforme; Brain Neoplasms, Malignant; Leptomeningeal Disease (LMD)
Keywords: glioblastoma; Ataxia-telangiectasia mutated kinase (ATM) inhibition; radiation therapy
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Meningeal Neoplasms; Hereditary Sensory and Autonomic Neuropathies; Inhibition, Psychological | interventions — Radiotherapy; AZD1390

STUDY DESIGN:
Intervention Model Description: AZD1390 will be administered to patients in three different Arms (A, B and C), with each arm receiving standard of care radiation therapy (RT) for their disease setting.
  In arms A and C, AZD1390 will be administered in three cycles: Cycle 0 (before RT), Cycle 1 (during RT) and Cycle 2 (after RT).
  In arm B, AZD1390 will be administered in cycle 1 only (during RT). Within each arm, AZD1390 will be administered in dose escalating cohorts, first in an intermittent and then in a consecutive fashion, to achieve daily administration prior to RT.
  **Arm B has now closed to recruitment**
  For Arm A, there is an optional food effect assessment during cycle 0. *Note: the food effect assessment is currently open to recruitment*
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: AZD1390 + Radiation Therapy (Experimental): AZD1390 administration plus 35 Gy of Intensity-modulated radiation therapy (IMRT) administered at daily fractions of 3.5 Gy over 10 fractions (2 weeks)
  Interventions: Radiation: Radiation Therapy; Drug: AZD1390
- Arm B: AZD1390 + Radiation Therapy (Experimental): AZD1390 administration plus 30 Gy of whole brain radiation therapy (WBRT) or partial brain radiation therapy (PBRT) administered at daily fractions of 3 Gy over 10 fractions (2 weeks).
  Interventions: Radiation: Radiation Therapy; Drug: AZD1390
- Arm C: AZD1390 + Radiation Therapy (Experimental): AZD1390 administration plus 60 Gy of intensity- modulated radiation therapy (IMRT) administered at daily fractions of 2 Gy over 30 fractions (6 weeks)
  Interventions: Radiation: Radiation Therapy; Drug: AZD1390

INTERVENTIONS:
Radiation: Radiation Therapy — 35 Gy of Intensity-modulated radiation therapy (IMRT) administered at daily fractions of 3.5 Gy over 10 fractions (2 weeks)
  Other Names: Radiotherapy; Radiation treatment; RT
  Arms: Arm A: AZD1390 + Radiation Therapy
Drug: AZD1390 — AZD1390 Administered in 3 Cycles depending on arm:
  Cycle 0: 1 dose prior to Radiation Therapy. Cycle 1: 2 weeks Intermittent or continuous dosing during Radiation Therapy. Cycle 2: 2 weeks adjuvant treatment after Radiation Therapy. For optional food effect assessment in Arm A, 2 doses prior to RT under both fed and fasted conditions. Note: the food effect assessment is currently open to recruitment.
  Arm A includes the Japan part following the same dosing administration.
  Other Names: ATM inhibitor
  Arms: Arm A: AZD1390 + Radiation Therapy
Radiation: Radiation Therapy — 30 Gy of whole brain radiation therapy (WBRT) or partial brain radiation therapy (PBRT) administered at daily fractions of 3 Gy over 10 fractions (2 weeks).
  Other Names: Radiotherapy; Radiation treatment; RT
  Arms: Arm B: AZD1390 + Radiation Therapy
Radiation: Radiation Therapy — 60 Gy of intensity- modulated radiation therapy (IMRT) administered at daily fractions of 2 Gy over 30 fractions (6 weeks)
  Other Names: Radiotherapy; Radiation treatment; RT
  Arms: Arm C: AZD1390 + Radiation Therapy
Drug: AZD1390 — AZD1390 administered in 1 Cycle. AZD1390 administration concomitantly with RT (2 weeks). Cycle 1 also contains an additional 5 days (post completion of RT with AZD1390 administration). Arm is Closed.
  Other Names: ATM inhibitor
  Arms: Arm B: AZD1390 + Radiation Therapy
Drug: AZD1390 — AZD1390 Administered in 3 Cycles depending on arm:
  Cycle 0: 1 dose prior to Radiation Therapy. Cycle 1: 6 weeks Intermittent or continuous dosing during Radiation Therapy. Cycle 2: 2 weeks adjuvant treatment after Radiation Therapy. Arm is closed.
  Other Names: ATM inhibitor
  Arms: Arm C: AZD1390 + Radiation Therapy

SUMMARY:
This study will test an investigational drug called AZD1390 in combination with radiation therapy for the treatment of brain tumors. This is the first time AZD1390 is being given to patients. This study will test safety, tolerability and PK (how the drug is absorbed, distributed and eliminated) of ascending doses of AZD1390 in combination with distinct regimens of radiation therapy

DETAILED DESCRIPTION:
This first time-in patients (FTIP), open-label, multicentre study of AZD1390 will be conducted in the United States, the United Kingdom and Japan. It consists of three treatment arms: Arm A, B, C. The Japan dose confirmation part (Japan part) is a sub-study of Arm A. Sites from Japan will only participate in the Japan part. This Phase 1 study will assess safety and tolerability of AZD1390 in combination with radiation therapy (RT) in brain malignancies. The combination cohorts have been designed to assess escalating cumulative doses of AZD1390 in settings with 3 different radiation treatment regimens:

* Arm A: 35 Gy over 2 weeks with intensity-modulated radiation therapy (IMRT) in patients with recurrent Glioblastoma Multiforme (GBM). Arm A will also include the food effect cohort
* Arms B: 30 Gy over two weeks with whole brain radiation therapy (WBRT)/ partial brain radiation therapy (PBRT) in patients with brain metastases. **Arm B has now closed to recruitment**
* Arm C: 60 Gy over 6 weeks (IMRT) in patients with primary GBM Each arm provides standard of care RT for the disease setting indicated with the experimental agent being administered in dose escalating cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Provision of formalin-fixed paraffin embedded tissue sample from primary or metastatic disease
* Karnofsky Performance Score of ≥60.
* Additional Inclusion Criteria Specific for Arm A and Japan:

  * Histologically proven diagnosis of GBM. Patients who have had RT for low-grade glioma (LGG) or grade 3 glioma and have subsequently relapsed to histologically confirmed GBM can be considered
  * A radiological diagnosis of recurrent/relapsed or progressive disease according to RANO criteria.
  * Completion of first-line radiation at least 6 months prior to Cycle 1 Day 1.
  * Patients with tumor-induced seizures must be well controlled on a stable anti-epileptic treatment
  * Willing to receive anti-epileptic prophylaxis for the duration of study drug administration.
* Additional Inclusion Criteria Specific for Arm B:

**Arm B has now closed to recruitment**

* Histologically proven diagnosis of solid tumor malignancy and Magnetic Resonance (MR) imaging documenting brain lesions.
* Not eligible for Stereotactic Radiosurgery (SRS) treatment of brain tumor.
* Patient has not received any previous brain RT to the area that is to be irradiated. Prior PBRT may be allowed if there is not significant overlap between the prior and new radiation fields.
* Non-CNS malignant disease must be sufficiently controlled so that patients can be without additional systemic therapy for the required washout period before starting therapy until 5 days after the end of RT. Required washout period before starting the first dose of AZD1390 (Cycle 1) is 28 days for immune checkpoint inhibitors and 7 days for all other agents
* Not received radiation to the lung fields within the past 8 weeks.
* No history of seizures related to the brain metastases or LMD.
* Receiving PBRT (rather than WBRT) during Cycle 1 as standard of care for brain metastases

  • Additional Inclusion Criteria Specific for Arm C:
* Histologically proven primary diagnosis of GBM with unmethylated O6-methylguanine-DNA methyltransferase (MGMT). Grade 4 astrocytoma or histology with molecular features of GBM can be considered.
* Determination of MGMT promoter status by methylation-specific polymerase chain reaction (PCR) or pyrosequencing per local institutional guidelines is required to assess eligibility for this Arm.
* Patients will have to undergo mutational testing for Isocitrate dehydrogenase 1 (IDH1) on a tumor specimen before entering study. Patients are eligible for Arm C regardless of their IDH1 mutational status.
* No history of uncontrolled seizures after surgery for primary GBM (despite adequate antiepileptic therapy) or with need for concurrent administration of more than 2 antiepileptic drugs.
* Willing to receive anti-epileptic prophylaxis for the duration of study drug administration

Additional Inclusion criteria for Food Effect Assessment (Arm A):

* For the fed assessment portion: fast overnight (for at least 10 hours) prior to consuming a high-fat meal consisting of approximately 800 to 1000 calories, with around 54% of the calories coming from fat.
* For the fasted assessment portion: fast overnight (for at least 10 hours prior to dosing) and until 4 hours after dosing.

*Note: the optional food effect assessment is currently open to enrolment*

Exclusion Criteria:

* Administration of chemotherapy or any investigational drug in the 28 days or carmustine (CCNU) or lomustine (BCNU) in the 6 weeks prior to receiving the first dose of treatment in Arms A and C. Administration of checkpoint inhibitors within 28 days prior to first dose of treatment and any other agent within 7 days of beginning study treatment in Arm B. Hormonal therapies are allowed during study treatment for patients in Arm B.
* History of severe brain-injury or stroke.
* Patient not eligible for sequential MRI evaluations are not eligible for this study.
* History of epileptic disorder or any seizure history unrelated to tumor
* Treatment with Strong inhibitors or inducers of CYP3A4 within 2 weeks prior to receiving study drug
* Concurrent therapy with other seizurogenic medications.
* Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
* Concurrent severe and/or uncontrolled medical condition (e.g., severe COPD).
* Prior treatment with pneumotoxic drugs, e.g. busulfan, bleomycin, within the past year. If prior therapy in lifetime, then excluded if history of pulmonary toxicities from administration. Patients who have received treatment with nitrosoureas (e.g., carmustine, lomustine) in the year before study entry without experiencing lung toxicity are allowed on study.
* History or presence of myopathy or raised creatine kinase (CK) >5 x upper limit of normal (ULN) on 2 occasions at screening.
* Cardiac dysfunction defined as: Myocardial infarction within six months of study entry, NYHA (New York Heart Association) Class II/III/IV heart failure, unstable angina, unstable cardiac arrhythmias
* Evidence of severe pulmonary infections, as judged by the investigator (For Japan part only this includes active infection including tuberculosis, chronic active or uncontrolled Hep B or Hep C)
* With the exception of alopecia, any unresolved toxicities from prior therapy greater than National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE 4.03) Grade 1 at the time of starting study treatment and patients with chronic Grade 2 unresolved toxicities may be eligible Additional exclusion criteria for Arm A and Japan Part
* Has previously received ATM inhibitor with concurrent RT

Additional Exclusion criteria for Food Effect Assessment (Arm A) (Not applicable for the Japan Part):

* Diabetes Type I, Type II, or steroid-induced diabetes.
* Undergoing systemic steroid treatment *Note: the food effect assessment is currently open to enrolment*

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-04-02 (Actual); Primary Completion 2026-09-16 (Estimated); Study Completion 2026-09-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | From the start of treatment until the end of the DLT period (approximately 6 weeks for Arm A, 3 weeks for Arm B and 10 weeks for Arm C)
  DLTs will be used to calculate the maximum tolerated dose (MTD). In each arm, the MTD of AZD1390 is the highest dose at which the predicted probability of a DLT is less than 25% in that specific RT setting
Incidence of adverse events (AEs) and serious adverse events (SAEs) | From the start of treatment until the end of the study (approximately 9 months after the last patient has started treatment)
  For each adverse event CTCAE grade and causality (related to AZD1390 or radiotherapy) will be collected.

SECONDARY OUTCOMES:
Event free survival (EFS) for Arms A and C only | From the start of treatment until the patient is off study (approximately 9 months after the last patient has started treatment)
  Defined as the time from the first dose of AZD1390 until the occurrence of any of the following events:
  1. Tumor progression or recurrence based on RANO criteria
  2. Secondary malignancy
  3. Change in tumor treatment due to increase clinical symptoms
  4. Death due to any cause
Objective response rate defined by RANO criteria for Arms A and C only | Every 8 weeks starting from 4 weeks after RT until the end of the study (approximately 9 months after the last patient has started treatment)
  The proportion of patients achieving a complete or partial tumor response (CR or PR) according to RANO criteria.
Objective response rate defined by RANO-BM criteria for Arm B only. **Arm B has now closed to recruitment** | From screening until the patient is off study, approximately 8 weeks
  The proportion of patients achieving a complete or partial tumor response (CR or PR) according to RANO-BM criteria.
Objective response rate defined by RECIST 1.1 criteria for Arm B only. **Arm B has now closed to recruitment** | From screening until the patient is off study, approximately 8 weeks
  The proportion of patients achieving a complete or partial tumor response (CR or PR) according to RECIST 1.1 criteria.
Maximum Observed Plasma Concentration (Cmax) of AZD1390 | At predefined intervals throughout the AZD1390 treatment period (approximately 5 weeks for Arm A, 2 weeks for Arm B and 9 weeks for Arm C)
  Blood samples will be collected to assess plasma concentrations of AZD1390 at a series of timepoints to derive Cmax
Time to observed Cmax (Tmax) for AZD1390 | At predefined intervals throughout the AZD1390 treatment period (approximately 5 weeks for Arm A, 2 weeks for Arm B and 9 weeks for Arm C)
  Blood samples will be collected to assess plasma concentrations of AZD1390 at a series of timepoints to derive Tmax
Area under the plasma concentration-time curve (AUC) for AZD1390 | At predefined intervals throughout the AZD1390 treatment period (approximately 5 weeks for Arm A, 2 weeks for Arm B and 9 weeks for Arm C)
  Blood samples will be collected to assess plasma concentrations of AZD1390 at a series of timepoints to derive AUC
Overall survival for Arms A and C only | From start of treatment until the patient dies, withdraws or the end of study is reached (approximately 9 months after the last patient has started treatment)
  Defined as the time from the first dose of AZD1390 until death from any cause
Assessment of the food effect of AZD1390 at the MTD for Arm A (if conducted) | At two predefined intervals during cycle 0 (at least 5 days apart)
  Blood samples will be collected to assess plasma concentrations of AZD1390 at a series of timepoints under fed and fasted conditions to derive Cmax, Tmax, and AUC

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wen, Principal Investigator — Dana-Farber Cancer Institute; Brandon Imber, Principal Investigator — Memorial Sloan Kettering Cancer Center; Mariza Daras, Principal Investigator — VCU Massey Cancer Center; Jan Drappatz, Principal Investigator — UPMC Hospital Radiation Oncology; Deborah Forst, Principal Investigator — Massachusetts General Hospital; Anthony Chalmers, Principal Investigator — Beatson West of Scotland Cancer Centre; Rajesh Jena, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust; Louise Murray, Principal Investigator — University of Leeds; Yoshitaka Narita, Principal Investigator — National Cancer Center Hospital; Yoshiki Arakawa, Principal Investigator — Kyoto University Hospital; Kazuhiko Mishima, Principal Investigator — Saitama Medical University International Medical Center
Locations (11):
- United States (4):
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Richmond, Virginia
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Hidaka-shi
  - Research Site, Kyoto
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, Glasgow
  - Research Site, Leeds
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home